CLINICAL TRIAL: NCT03083197
Title: The Scrub Typhus Antibiotic Resistance Trial (START) Comparing Doxycycline and Azithromycin Treatment Modalities in Areas of Reported Antimicrobial Resistance for Scrub Typhus
Brief Title: Scrub Typhus Antibiotic Resistance Trial
Acronym: START
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Shoklo Malaria Research Unit (Other); Chiangrai Prachanukroh Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: START
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Scrub Typhus
Keywords: Scrub Typhus; Antibiotic Resistance
MeSH Terms: conditions — Scrub Typhus | interventions — Doxycycline; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Doxycycline 7 days (Active Comparator): loading dose 200mg PO, then 100mg PO every 12 hours for 7 days
  Interventions: Drug: Doxycycline 7 days
- Doxycycline 3 days (Active Comparator): loading dose 200mg PO, then 100mg PO every 12 hours for 3 days
  Interventions: Drug: Doxycycline 3 days
- Azithromycin 3 days (Active Comparator): loading dose 1000mg PO on day 1, then 500mg PO every 24 hours on days 2 and 3
  Interventions: Drug: Azithromycin 3 days

INTERVENTIONS:
Drug: Doxycycline 7 days — loading dose 200mg PO, then 100mg PO every 12 hours for 7 days
  Arms: Doxycycline 7 days
Drug: Doxycycline 3 days — loading dose 200mg PO, then 100mg PO every 12 hours for 3 days
  Arms: Doxycycline 3 days
Drug: Azithromycin 3 days — loading dose 1000mg PO on day 1, then 500mg PO every 24 hours on days 2 and 3
  Arms: Azithromycin 3 days

SUMMARY:
Study type: Randomized Control Treatment Trial

Study population: Male and female patients with ≥15 years of age and acute scrub typhus

Duration: 2 years

Study Design: Prospective, open-label, randomized-controlled treatment trial in patients ≥15 years old admitted to hospital with acute scrub typhus. Randomization into 3 oral treatment arms (each n=59 patients, total n=177): i) 7 days of doxycycline, ii) 3 days of doxycycline, and iii) 3 days of azithromycin

Primary Objective: To evaluate the clinical and microbiological responses in scrub typhus patients to three oral treatment regimens: 7 days of doxycycline, 3 days of doxycycline, and 3 days of azithromycin

Secondary Objectives:

1. To perform pharmacokinetic/pharmacodynamics (PK/PD) characterization of the therapeutic responses for doxycycline and azithromycin, incl. serial bacterial load measurements.
2. To define clinical, bacterial, pathophysiological and pharmacological factors associated with disease severity, fever-clearance times (FCT), treatment failures and relapse/re-infection.
3. To determine the minimum inhibitory concentrations (MIC) of clinical Orientia tsutsugamushi isolates to doxycycline, azithromycin and chloramphenicol, using in vitro growth-inhibition assays
4. To genotype all clinical isolates using whole genome sequencing for comparative genomics.
5. To dissect the natural immune response in scrub typhus, using antigen-specific cellular immune and antibody studies, and cytokine profiling

DETAILED DESCRIPTION:
The funder is USAMRMC - MIDRP and Grant No. DHP-Award D6.7_15_C2_I_15_J9_1317

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years old
* Hospitalization with acute undifferentiated fever (temperature > 37.5°C, tympanic) ≤14 days or patients admitted to hospital with a history of fever ≤ 14 days who subsequently develop fever within 24 hours of admission
* Clinically suspected scrub typhus: defined as acute undifferentiated fever with no clear focus of infection and negative malaria blood smear and/or negative malaria RDT. Patients may have one, none, or a combination of other clinical findings such as eschar, rash, lymphadenopathy, headache, myalgia, cough, nausea and abdominal discomfort.
* A positive scrub typhus RDT (Scrub Typhus IgM RDT, InBios International, Seattle, WA, USA) and/or positive PCR-based detection of O. tsutsugamushi DNA from the admission blood sample
* Written informed consent and/or, written informed assent as required
* Able to take oral medication

Exclusion Criteria:

* Known hypersensitivity to tetracycline, doxycycline or azithromycin
* Administration of doxycycline, azithromycin, chloramphenicol, rifampicin, or tetracycline during the preceding 7 days
* Pregnancy or breast-feeding
* Patients with myasthenia gravis or systemic lupus erythematosus
* Patients with an established infection (diagnostic test required) e.g. acute malaria, dengue, leptospirosis, typhoid, Japanese encephalitis etc.
* Current TB or TB treatment in ≤ 6 months (contain active antibiotics against Orientia spp.)
* Current HAART use for HIV, long term use of immunosuppressants (e.g. steroids, chemotherapy, TNF-inhibitors and related agents)
* Patients with severe disease whom the clinical team feel their condition necessitates the need for additional scrub typhus treatment beyond the allocated antibiotic treatment assigned at randomization (e.g. IV chloramphenicol and/or PO/NG rifampicin)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Fever clearance time (FCT) | at least 24 hours
  Based on the time from first dose of antibiotic treatment to when the tympanic temperature first falls ≤37.5°C and remains ≤37.5°C for at least 24 hours, outside of the influence of paracetamol.

SECONDARY OUTCOMES:
Resolution of bacteraemia in relation to Drug plasma level | 8 Weeks
Occurrence of severe disease or treatment failure/relapse | 8 Weeks
Presence of in vitro antimicrobial resistance | 8 Weeks
  (Minimum inhibitory concentrations (MIC) over susceptibility cut off)
Genotyping of clinical Orientia tsutsugamushi isolates (56kDa gene +/- whole genome sequencing) | 2 years
  Genotyping of clinical OT isolates will be performed on patient samples that are PCR positive (approximately 50-60%) and/or culture positive (approximately 30%). Extracted DNA will be sent for 56kDa gene sequencing +/- whole genome sequencing, revealing the clinically important strains and allowing for comparative analysis with disease severity and patient outcomes.
Antigen-specific positive cellular and humoral immune responses | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Daniel Paris, Principal Investigator — Mahidol-Oxford Tropical Medicine Research Unit, Bangkok, Thailand
Locations (2):
- Thailand (2):
  - Shoklo-Malaria Research Unit (SMRU), Mae Sot, Changwat Tak
  - Chiangrai Prachanukroh Hospital, Chiang Rai

IPD SHARING:
Plan to Share IPD: Undecided